CLINICAL TRIAL: NCT00466050
Title: Correlation Between Serum Markers of Unstable Plaque and Virtual Histology of Unstable Plaque Visualized by IVUS
Acronym: IVUS
Status: Completed | Type: Observational
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Ziv Hospital, Ziv Hospital
Other Study IDs: HP-7-234-S
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2007-04

CONDITIONS: Acute Coronary Thrombose; Plaque Rupture; Acute Coronary Syndrome
Keywords: plaque rupture,; acute coronary thrombose,; coronary angiography,; IVUS
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Thirty patients scheduled to coronary angiography and IVUS in according to their treating physician decision will be enrolled in the study. The coronary angiography and IVUS will be done on according to regular clinical standards.

As the study protocol, 40 cc of blood will be drawn from the patients after written informed consent.

The laboratory tests will be processed for the above mentioned serum markers of unstable plaque.

A multivariate correlation test will be done between the different serum markers and the plaque morphology by angiography and composition (virtual histology) by IVUS.

DETAILED DESCRIPTION:
Serum markers of unstable plaque Myeloperoxidase is a lysosomal enzyme, requiring heme as a cofactor, released from neutrophilic granules, monocytes, and some subtypes of tissue macrophages.

Myeloperoxidase is also linked to oxidation of lipids in low-density lipoproteins (LDL), dysfunctional high density lipoproteins (HDL), and consumption of nitric oxide thereby rendering the normally anti-thrombotic endothelial surface thrombogenic via the expression of various pro-thrombotic and anti-fibrinolytic factor (19).

Myeloperoxidase plays a role in the degradation of the fibrous cap, making it both a marker of inflammation and one of plaque instability.

Interest in MPO intensified after a report by Brennan and colleagues (20) indicated that a single initial measurement of plasma myeloperoxidase independently predicts the early risk of myocardial infraction, as well as the risk of major adverse cardiac events in the ensuring 30-day and 6-month periods.

Two markers of recent interest relating to plaque vulnerability pregnancy-associated protein A(PAPP-A) and placenta growth factor (P1GF).

Pregnancy -associated protein A is a metalloproteinase, initially identified in the sera of pregnant women (21).

A large study has illustrated that decreases in IGF-1 appear to be cardio protective, yet some research shows that increases in PAPP-A, which should also increase the bioavailability of IGF-1, may be a relevant marker for the presence and extent of coronary atherosclerosis (22). It is believed that PAPP-A is released during plaque destabilization and appears to be a valuable indicator of unstable angina and acute MI in patients lacking other indicators of necrosis (23).

Placenta growth factor, is a member of the vascular endothelial growth factor family, which stimulates vascular smooth muscle growth, recruits macrophages into atherosclerotic lesion, up-regulates production of tumor necrosis factor- and monocyte chemotactic protein 1 by macrophages, and stimulates pathological angiogenesis (24). It appears to be an initiator of the inflammatory process.

In one study, elevated P1GF levels not only identified patients with acute chest pain who developed ACS, but also those patients with an increased risk of recurrent instability after hospital discharge (25).

Plasma elevation of CRP have been reported fraction, and are acute ischemia and myocardial in fraction, and are predictive of the risk of recurrent ischemia among hospitalization patients with unstable angina (26).

Matrix metalloproteinases. MMPs are a diverse family of powerful, zinc-containing enzymes expressed by macrophage- derived foam cells, SMCs and other vascular cells within atherosclerotic lesions (27) .It has been previously demonstrated that MMPs are responsible for remodeling of the ECM during all stages of atheromatous development and may directly contribute to fibrous cap weakening and plaque rupture within disease arteries (28).

CD40 ligand (CD40L) is an immunoregulatory transmembrane protein that belongs to the tumor necrosis factor (TNF) super family. It is expressed on the surface of many cells types, including leukocytes, ECs, SMSs, macrophages, and activated platelets (29). Ligand receptor binding on these cells triggers the expression and secretion of a variety of pro-inflammatory and procoagulant mediators, including CAMs, cytokines, chemokines, growth factors, MMPs, and TF (29). Recent data suggest that CD40L plays a central role in the inflammatory process that contributes to plaque destabilization in CAD (30), and elevation in soluble, biologically active CD40L (Scd40l) have been demonstrated in the serum of ACS patients (31).

Paraoxonase and atherogenic HDL The enzyme PON1 is known to be tightly bound with HDL in serum, and several studies suggest that it is this association that contributes to the protection conferred by HDL against LDL oxidation (33-36).

The aim of the study is to find a correlation between serum markers of unstable plaque and virtual histology of unstable plaque visualized by IVUS.

Patients and methods:

Thirty patients scheduled to coronary angiography and IVUS in according to their treating physician decision will be enrolled in the study. The coronary angiography and IVUS will be done on according to regular clinical standards.

As the study protocol, 40 cc of blood will be drawn from the patients after written informed consent.

The laboratory tests will be processed for the above mentioned serum markers of unstable plaque.

A multivariate correlation test will be done between the different serum markers and the plaque morphology by angiography and composition (virtual histology) by IVUS.

ELIGIBILITY:
Inclusion Criteria:

* Both genders: males and females
* Age - above 18 years
* Patients scheduled to coronary angiography and IVUS
* Written Informed Consent Form

Exclusion Criteria:

* Pregnant or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to coronary angiography and IVUS
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2007-04; Primary Completion 2008-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Osamah Hussein, MD, Principal Investigator — Ziv Medical Center; Alon Marmor, Prof, Principal Investigator — Ziv Medical Center
Locations (1):
- Heart Institute ,Ziv Medical Center, Safed, Israel

REFERENCES:
- [Background] Davies MJ, Thomas AC. Plaque fissuring--the cause of acute myocardial infarction, sudden ischaemic death, and crescendo angina. Br Heart J. 1985 Apr;53(4):363-73. doi: 10.1136/hrt.53.4.363. No abstract available. PMID 3885978
- [Background] Virmani R, Kolodgie FD, Burke AP, Farb A, Schwartz SM. Lessons from sudden coronary death: a comprehensive morphological classification scheme for atherosclerotic lesions. Arterioscler Thromb Vasc Biol. 2000 May;20(5):1262-75. doi: 10.1161/01.atv.20.5.1262. No abstract available. PMID 10807742
- [Background] Frink RJ. Chronic ulcerated plaques: new insights into the pathogenesis of acute coronary disease. J Invasive Cardiol. 1994 Jun;6(5):173-85. PMID 10155066
- [Background] Mann J, Davies MJ. Mechanisms of progression in native coronary artery disease: role of healed plaque disruption. Heart. 1999 Sep;82(3):265-8. doi: 10.1136/hrt.82.3.265. PMID 10455072
- [Background] Falk E, Shah PK, Fuster V. Coronary plaque disruption. Circulation. 1995 Aug 1;92(3):657-71. doi: 10.1161/01.cir.92.3.657. No abstract available. PMID 7634481
- [Background] Schmermund A, Erbel R. Unstable coronary plaque and its relation to coronary calcium. Circulation. 2001 Oct 2;104(14):1682-7. doi: 10.1161/hc3901.093339. PMID 11581149
- [Background] Giroud D, Li JM, Urban P, Meier B, Rutishauer W. Relation of the site of acute myocardial infarction to the most severe coronary arterial stenosis at prior angiography. Am J Cardiol. 1992 Mar 15;69(8):729-32. doi: 10.1016/0002-9149(92)90495-k. PMID 1546645
- [Background] Nobuyoshi M, Tanaka M, Nosaka H, Kimura T, Yokoi H, Hamasaki N, Kim K, Shindo T, Kimura K. Progression of coronary atherosclerosis: is coronary spasm related to progression? J Am Coll Cardiol. 1991 Oct;18(4):904-10. doi: 10.1016/0735-1097(91)90745-u. PMID 1894863
- [Background] Klingensmith JD, Vince DG, Kuban BD, Shekhar R, Tuzcu EM, Nissen SE, Cornhill JF. Assessment of coronary compensatory enlargement by three-dimensional intravascular ultrasound. Int J Card Imaging. 2000 Apr;16(2):87-98. doi: 10.1023/a:1006333619358. PMID 10928343
- [Background] Nissen SE, Gurley JC, Grines CL, Booth DC, McClure R, Berk M, Fischer C, DeMaria AN. Intravascular ultrasound assessment of lumen size and wall morphology in normal subjects and patients with coronary artery disease. Circulation. 1991 Sep;84(3):1087-99. doi: 10.1161/01.cir.84.3.1087. PMID 1884441
- [Background] Schoenhagen P, Ziada KM, Kapadia SR, Crowe TD, Nissen SE, Tuzcu EM. Extent and direction of arterial remodeling in stable versus unstable coronary syndromes : an intravascular ultrasound study. Circulation. 2000 Feb 15;101(6):598-603. doi: 10.1161/01.cir.101.6.598. PMID 10673250
- [Background] Tuzcu EM, Hobbs RE, Rincon G, Bott-Silverman C, De Franco AC, Robinson K, McCarthy PM, Stewart RW, Guyer S, Nissen SE. Occult and frequent transmission of atherosclerotic coronary disease with cardiac transplantation. Insights from intravascular ultrasound. Circulation. 1995 Mar 15;91(6):1706-13. doi: 10.1161/01.cir.91.6.1706. PMID 7882477
- [Background] von Birgelen C, de Vrey EA, Mintz GS, Nicosia A, Bruining N, Li W, Slager CJ, Roelandt JR, Serruys PW, de Feyter PJ. ECG-gated three-dimensional intravascular ultrasound: feasibility and reproducibility of the automated analysis of coronary lumen and atherosclerotic plaque dimensions in humans. Circulation. 1997 Nov 4;96(9):2944-52. doi: 10.1161/01.cir.96.9.2944. PMID 9386161
- [Background] Palmer ND, Northridge D, Lessells A, McDicken WN, Fox KA. In vitro analysis of coronary atheromatous lesions by intravascular ultrasound; reproducibility and histological correlation of lesion morphology. Eur Heart J. 1999 Dec;20(23):1701-6. doi: 10.1053/euhj.1999.1627. PMID 10562477
- [Background] Thieme T, Wernecke KD, Meyer R, Brandenstein E, Habedank D, Hinz A, Felix SB, Baumann G, Kleber FX. Angioscopic evaluation of atherosclerotic plaques: validation by histomorphologic analysis and association with stable and unstable coronary syndromes. J Am Coll Cardiol. 1996 Jul;28(1):1-6. doi: 10.1016/0735-1097(96)00108-8. PMID 8752786
- [Background] Waxman S, Sassower MA, Mittleman MA, Zarich S, Miyamoto A, Manzo KS, Muller JE, Abela GS, Nesto RW. Angioscopic predictors of early adverse outcome after coronary angioplasty in patients with unstable angina and non-Q-wave myocardial infarction. Circulation. 1996 Jun 15;93(12):2106-13. doi: 10.1161/01.cir.93.12.2106. PMID 8925578
- [Background] Nicholls SJ, Hazen SL. Myeloperoxidase and cardiovascular disease. Arterioscler Thromb Vasc Biol. 2005 Jun;25(6):1102-11. doi: 10.1161/01.ATV.0000163262.83456.6d. Epub 2005 Mar 24. PMID 15790935
- [Background] Brennan ML, Penn MS, Van Lente F, Nambi V, Shishehbor MH, Aviles RJ, Goormastic M, Pepoy ML, McErlean ES, Topol EJ, Nissen SE, Hazen SL. Prognostic value of myeloperoxidase in patients with chest pain. N Engl J Med. 2003 Oct 23;349(17):1595-604. doi: 10.1056/NEJMoa035003. PMID 14573731
- [Background] Wald NJ, George L, Smith D, Densem JW, Petterson K. Serum screening for Down's syndrome between 8 and 14 weeks of pregnancy. International Prenatal Screening Research Group. Br J Obstet Gynaecol. 1996 May;103(5):407-12. doi: 10.1111/j.1471-0528.1996.tb09765.x. PMID 8624312
- [Background] Cosin-Sales J, Kaski JC, Christiansen M, Kaminski P, Oxvig C, Overgaard MT, Cole D, Holt DW. Relationship among pregnancy associated plasma protein-A levels, clinical characteristics, and coronary artery disease extent in patients with chronic stable angina pectoris. Eur Heart J. 2005 Oct;26(20):2093-8. doi: 10.1093/eurheartj/ehi433. Epub 2005 Jul 29. PMID 16055491
- [Background] Bayes-Genis A, Conover CA, Overgaard MT, Bailey KR, Christiansen M, Holmes DR Jr, Virmani R, Oxvig C, Schwartz RS. Pregnancy-associated plasma protein A as a marker of acute coronary syndromes. N Engl J Med. 2001 Oct 4;345(14):1022-9. doi: 10.1056/NEJMoa003147. PMID 11586954
- [Background] Autiero M, Luttun A, Tjwa M, Carmeliet P. Placental growth factor and its receptor, vascular endothelial growth factor receptor-1: novel targets for stimulation of ischemic tissue revascularization and inhibition of angiogenic and inflammatory disorders. J Thromb Haemost. 2003 Jul;1(7):1356-70. doi: 10.1046/j.1538-7836.2003.00263.x. PMID 12871269
- [Background] Heeschen C, Dimmeler S, Fichtlscherer S, Hamm CW, Berger J, Simoons ML, Zeiher AM; CAPTURE Investigators. Prognostic value of placental growth factor in patients with acute chest pain. JAMA. 2004 Jan 28;291(4):435-41. doi: 10.1001/jama.291.4.435. PMID 14747500
- [Background] Liuzzo G, Biasucci LM, Gallimore JR, Grillo RL, Rebuzzi AG, Pepys MB, Maseri A. The prognostic value of C-reactive protein and serum amyloid a protein in severe unstable angina. N Engl J Med. 1994 Aug 18;331(7):417-24. doi: 10.1056/NEJM199408183310701. PMID 7880233
- [Background] Galis ZS, Sukhova GK, Kranzhofer R, Clark S, Libby P. Macrophage foam cells from experimental atheroma constitutively produce matrix-degrading proteinases. Proc Natl Acad Sci U S A. 1995 Jan 17;92(2):402-6. doi: 10.1073/pnas.92.2.402. PMID 7831299
- [Background] Lendon CL, Davies MJ, Born GV, Richardson PD. Atherosclerotic plaque caps are locally weakened when macrophages density is increased. Atherosclerosis. 1991 Mar;87(1):87-90. doi: 10.1016/0021-9150(91)90235-u. PMID 1872926
- [Background] Henn V, Slupsky JR, Grafe M, Anagnostopoulos I, Forster R, Muller-Berghaus G, Kroczek RA. CD40 ligand on activated platelets triggers an inflammatory reaction of endothelial cells. Nature. 1998 Feb 5;391(6667):591-4. doi: 10.1038/35393. PMID 9468137
- [Background] Mach F, Schonbeck U, Sukhova GK, Atkinson E, Libby P. Reduction of atherosclerosis in mice by inhibition of CD40 signalling. Nature. 1998 Jul 9;394(6689):200-3. doi: 10.1038/28204. PMID 9671306
- [Background] Heeschen C, Dimmeler S, Hamm CW, van den Brand MJ, Boersma E, Zeiher AM, Simoons ML; CAPTURE Study Investigators. Soluble CD40 ligand in acute coronary syndromes. N Engl J Med. 2003 Mar 20;348(12):1104-11. doi: 10.1056/NEJMoa022600. PMID 12646667
- [Background] Ueda Y, Asakura M, Hirayama A, Komamura K, Hori M, Komada K. Intracoronary morphology of culprit lesions after reperfusion in acute myocardial infarction: serial angioscopic observations. J Am Coll Cardiol. 1996 Mar 1;27(3):606-10. doi: 10.1016/0735-1097(95)00534-x. PMID 8606271
- [Background] Mackness MI, Arrol S, Durrington PN. Paraoxonase prevents accumulation of lipoperoxides in low-density lipoprotein. FEBS Lett. 1991 Jul 29;286(1-2):152-4. doi: 10.1016/0014-5793(91)80962-3. PMID 1650712
- [Background] Mackness MI, Arrol S, Abbott C, Durrington PN. Protection of low-density lipoprotein against oxidative modification by high-density lipoprotein associated paraoxonase. Atherosclerosis. 1993 Dec;104(1-2):129-35. doi: 10.1016/0021-9150(93)90183-u. PMID 8141836
- [Background] Mackness MI, Abbott C, Arrol S, Durrington PN. The role of high-density lipoprotein and lipid-soluble antioxidant vitamins in inhibiting low-density lipoprotein oxidation. Biochem J. 1993 Sep 15;294 ( Pt 3)(Pt 3):829-34. doi: 10.1042/bj2940829. PMID 8379937
- [Background] Mackness MI, Durrington PN. HDL, its enzymes and its potential to influence lipid peroxidation. Atherosclerosis. 1995 Jun;115(2):243-53. doi: 10.1016/0021-9150(94)05524-m. PMID 7661883